CLINICAL TRIAL: NCT01306578
Title: Comparison of Intravenous Immunoglobulin and Plasma Exchange in Treatment of Mechanically Ventilated Children With Guillain Barre Syndrome. A Randomized Study.
Brief Title: Intravenous Immunoglobulin (IVIG) Versus Plasma Exchange (PE) for Ventilated Children With Guillain Barre Syndrome (GBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Dr. Mohammed El-Bayoumi, MD, FRCPCH, Head of PICU - Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUCH-GBS
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Guillain Barre Syndrome
Keywords: Guillain Barre syndrome; IVIG; Plasma exchange
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Immunoglobulins, Intravenous; Plasma Exchange; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG group (Active Comparator): 20 children randomized to receive IVIG for 5 days at a dose of 0.4 g/kg/day
  Interventions: Drug: IVIG
- Plasma Exchange (Active Comparator): 21 children randomized to receive 5 sessions of 1 volume plasma exchange per day for 5 consecutive days
  Interventions: Procedure: Plasma Exchange

INTERVENTIONS:
Drug: IVIG — Intravenous Immune Globulin at a dose 0f 0.4 g/kg/day for 5 consecutive days
  Other Names: Sandglobin
  Arms: IVIG group
Procedure: Plasma Exchange — Five sessions of plasma exchange, single plasma volume each, for 5 consecutive days
  Other Names: Plasmapheresis
  Arms: Plasma Exchange

SUMMARY:
Comparing whether intravenous immune globulin or plasma exchange is superior in treating mechanically ventilated children with Guillain Barre syndrome.

DETAILED DESCRIPTION:
Children with Guillain Barre syndrome (GBS) admitted to PICU at Mansoura University Children Hospital, Mansoura, Egypt with the need for mechanical ventilation were prospectively enrolled in the study.

Cases were diagnosed according to clinical criteria. The decisions to initiate, wean and terminate mechanical ventilation were made independently by the attending consultant in accordance with the unit guidelines.

Outcome variables measured were duration of mechanical ventilation, length of PICU stay and ability to walk unaided 4 weeks after PICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age: children from 1 month - 18 years old
* Clinical diagnosis of Guillain Barre syndrome
* Requirement of mechanical ventilation

Exclusion Criteria:

* Need for mechanical ventilation beyond 14 days from disease onset
* Child receiving IVIG or PE prior to enrollment

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 21 days (average)
  How many days did the mechanical ventilation continue

SECONDARY OUTCOMES:
PICU stay | 28 days (average)
  How many days did the child spend on PICU
Ability to walk | 4 weeks from PICU discharge
  Ability of the child to walk unaided at 4 weeks from PICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A El-Bayoumi, MD, FRCPCH, Principal Investigator — Head of PICU, Mansoura University Children Hospital
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Derived] Saleh M, Boukhdoud M, Boukhdoud H, Al Zein M, Salameh P. Landscape of Guillain-Barre Syndrome Interventional Clinical Trials. J Clin Neuromuscul Dis. 2023 Mar 1;24(3):119-129. doi: 10.1097/CND.0000000000000441. PMID 36809199
- [Derived] El-Bayoumi MA, El-Refaey AM, Abdelkader AM, El-Assmy MM, Alwakeel AA, El-Tahan HM. Comparison of intravenous immunoglobulin and plasma exchange in treatment of mechanically ventilated children with Guillain Barre syndrome: a randomized study. Crit Care. 2011 Jul 11;15(4):R164. doi: 10.1186/cc10305. PMID 21745374